CLINICAL TRIAL: NCT01359046
Title: Randomized Control Trial of Silver-alloy Impregnated Suprapubic Catheters in Urogynecology Patients
Brief Title: Silver-impregnated Suprapubic Catheters (SPC) in Urogynecology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John B. Gebhart, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10-007421
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-04

CONDITIONS: Infection Associated With Catheter; Urinary Tract Infection
Keywords: CAUTI; UTI
MeSH Terms: conditions — Catheter-Related Infections; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- silver SPC (Experimental): Subjects randomized to receive silver-impregnated SPC.
  Interventions: Device: silver SPC
- standard SPC (Active Comparator): subjects randomized to receive standard SPC.
  Interventions: Device: standard SPC

INTERVENTIONS:
Device: silver SPC — subject randomized to receive silver alloy impregnated catheter
  Arms: silver SPC
Device: standard SPC — subject randomized to receive standard catheter
  Arms: standard SPC

SUMMARY:
The purpose of this study is to compare urinary tract infection rates among women undergoing urogynecological procedures with a silver-alloy suprapubic catheter compared to the standard suprapubic catheter.

DETAILED DESCRIPTION:
Urinary catheters are used routinely in the postoperative care of urogynecology patients after surgery involving the genitourinary tract. However, Urinary tract infections(UTI) associated with indwelling catheter is the second leading cause of nosocomial infections. 20% of hospital acquired bacteremia arise from UTI with an associated mortality of 10%.

There are many different types of catheters available for use. Standard indwelling catheters are made from a variety of materials including polyvinyl chlorine, plastic, plain latex, polytetrafluoroethylene, silicone elastomer, pure silicone hydrogel and polymer hydromer. Specialized catheters have been developed with the aim of reducing infection. Strategies generally involved coating the inner, outer or both surfaces of the catheter with antimicrobial materials. These materials can be antibiotic or antiseptic with the most common antiseptic material used being silver. Silver ions are bactericidal, are used safely when applied topically to humans and used in controlling infections.

Previous studies comparing UTI rates in transurethral catheters have reported a significant reduction of UTI rate in silver-alloy catheters with a range of 5-12% compared to standard catheters with a range of 7-50%. There are no studies comparing the UTI rate in silver-alloy supra-pubic catheters to standard supra-pubic catheters. The investigators hypothesize that this study will show a statistically significant decrease in UTI rate among the individuals with a silver-alloy suprapubic catheter compared to the standard silver-alloy catheter.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring intra-operative placement of suprapubic catheters as part of routine post-operative care for repair of vaginal anterior compartment prolapse i.e. patients undergoing anterior colporrhaphy, Burch colposuspension, with or without mid-urethral sling

Exclusion Criteria:

* Known UTI at time of surgery
* Unable to provide informed consent
* Use of chronic intermittent self-catheterization pre-operatively
* Use of chronic prophylactic antibiotics
* Use of antibiotics for any indication other than UTI during peri-operative and 6-week post-operative period
* Presence of fistula involving urogenital tract
* Use of chronic steroids or immunosuppressant
* Immunocompromised patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2011-07; Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Gebhart, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Singh R, Hokenstad ED, Wiest SR, Kim-Fine S, Weaver AL, McGree ME, Klingele CJ, Trabuco EC, Gebhart JB. Randomized controlled trial of silver-alloy-impregnated suprapubic catheters versus standard suprapubic catheters in assessing urinary tract infection rates in urogynecology patients. Int Urogynecol J. 2019 May;30(5):779-787. doi: 10.1007/s00192-018-3726-z. Epub 2018 Aug 25. PMID 30145671
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Silver SPC | Standard SPC
Started | 144 | 144
Completed | 137 | 127
Not Completed | 7 | 17
Not completed — Did not receive allocated intervention | 6 | 6
Not completed — Physician Decision | 1 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Silver SPC | Standard SPC | Total
Number analyzed (Participants) | 137 | 127 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.5) | 66.3 (10.4) | 65.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 127 | 264
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 131 | 124 | 255
  Non-white | 5 | 2 | 7
  Unknown | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 137 | 127 | 264
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (5.0) | 27.8 (5.2) | 27.7 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Urinary Tract Infection Rate
Description: Number of subjects diagnosed with a urinary tract infection (UTI) within 6 weeks of surgery. A UTI is defined as any symptoms requiring antibiotic treatment, a urine culture with >10^5 cfu/mL, or a urine culture with >10^3 cfu/mL and evidence of pyuria.
Time Frame: within 6 weeks post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Silver SPC | Standard SPC
Number analyzed (Participants) | 131 | 123
Participants | 24 | 29
Statistical Analysis 1: Comparison: Silver SPC vs Standard SPC; Test type: Superiority; p = 0.30, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Risk of Urinary Tract Infections in Diabetics
Description: Number of diabetic subjects diagnosed with a urinary tract infection within 6 weeks post surgery.
Time Frame: within 6 weeks post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Silver SPC | Standard SPC
Number analyzed (Participants) | 15 | 16
Participants | 4 | 8
Statistical Analysis 1: Comparison: Silver SPC vs Standard SPC; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were captured and reported from enrollment to the 6 week post-operative period, which is the end of study treatment follow-up.
Arm/Group | Silver SPC | Standard SPC
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/127
Serious Adverse Events (participants affected / at risk) | 3/137 | 3/127
Other Adverse Events (participants affected / at risk) | 0/137 | 0/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silver SPC (N=137) | Standard SPC (N=127)
Reoperation (Surgical and medical procedures) | 1 (1) | 1 (1)
Pulmonary embolism (General disorders) | 0 (0) | 1 (1)
Ureteral stent placement (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Hernaturia (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-02-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT01359046/Prot_SAP_000.pdf